CLINICAL TRIAL: NCT03554551
Title: Imaging the Vesicular Acetylcholine Transporter Using 18Fluoro-fluoroethoxybenzovesamicol (18F-FEOBV) Positron Emission Tomography(PET) in Parkinsons Disease
Brief Title: Imaging the Vesicular Acetylcholine Transporter Using 18F-FEOBV PET in Parkinsons Disease
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Jacob Horsager, Principal investigator, Aarhus University Hospital
Other Study IDs: FEO-PD
Record Dates: First submitted 2018-05-31; First posted 2018-06-13 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Parkinson Disease
Keywords: Parasympathetic
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with Parkinsons disease: Disease duration > 4 years, Hoehn & Yahr stage 2-3, 50-85 years old
- Healthy controls: 50-85 years

SUMMARY:
Patients with Parkinson's disease (PD) often display symptoms, such as constipation, due to denervation of the cholinergic nerves in the gut. It has been hypothesized that PD initiates in the gut years prior to diagnosis. To gain a detailed understanding of the early stages of PD, techniques for quantification of cholinergic nerves are needed. The PET tracer 18F-FEOBV binds specifically to the vesicular acetylcholine transporter, situated in presynaptic cholinergic nerve terminals. The investigators will investigate 18F-FEOBV uptake in the brain and internal organs of 15 patients with moderate-stage PD and compare to 15 healthy controls. Furthermore, findings are correlated to validated clinical tests of the autonomic nervous system. The aim is to validate 18F-FEOBV PET/CT as a clinical imaging modality to diagnose parasympathetic denervation in PD.

ELIGIBILITY:
Inclusion Criteria:

* Parkinsons disease, disease duration > 4 years, Hoehn & Yahr stage 2-3

Exclusion Criteria:

* Significant neurological diseases (e.g. stroke, tumor)
* Significant psychiatric disease
* Previous major surgery on thoracic and/or abdominal organs
* Significant medical disease (e.g. heart- or liver failure)
* Inflammatory bowel disease
* Gluten intolerance
* Diabetes
* Magnetic Resonance (MR) contraindications (metal in body, claustrophobia)
* Allergy to CT-contrast fluid
* Pacemaker
* Any current or previous cancer involving internal organs
* Peripheral neuropathy (except Parkinsons disease related)

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parkinson patients are moderate stage disease. Healthy subjects have to meet the criteria below.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2018-08-08 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

PRIMARY OUTCOMES:
Density of vesicular acetylcholine transporter | Day 1
  Average density will be determined in each group for intestine, pancreas, suprarenal gland, heart and relevant areas of the brain. Group differences will be calculated

SECONDARY OUTCOMES:
Correlation to measurements of gastrointestinal denervation | Day 1
  Density of vesicular acetylcholine transporter will be correlated to symptoms of gastrointestinal autonomic denervation (constipation, gastroparesis).
Correlation to measurements of dysautonomia | Day 1
  Density of vesicular acetylcholine transporter will be correlated to measurements of dysautonomia (orthostatic hypotension, colon transit time)
Correlation to measurements of neuropsychological tests | Day 1
  Cerebral density of vesicular acetylcholine transporter is correlated with neuropsychological test scores.

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Region Midt, Denmark

REFERENCES:
- [Derived] Horsager J, Okkels N, Van Den Berge N, Jacobsen J, Schact A, Munk OL, Vang K, Bender D, Brooks DJ, Borghammer P. In vivo vesicular acetylcholine transporter density in human peripheral organs: an [18F]FEOBV PET/CT study. EJNMMI Res. 2022 Apr 1;12(1):17. doi: 10.1186/s13550-022-00889-9. PMID 35362761